CLINICAL TRIAL: NCT03853876
Title: A Natural History Study of Aspartylglucosaminuria
Acronym: AGU
Status: Terminated | Type: Observational
Why Stopped: Discontinued AGU development program
Sponsor: Neurogene Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AGU-100
Record Dates: First submitted 2019-01-17; First posted 2019-02-26 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Aspartylglucosaminuria; Aspartylglucosamidase (AGA) Deficiency; Lysosomal Storage Diseases
MeSH Terms: conditions — Aspartylglucosaminuria; Aspartylglucosamidase (AGA) deficiency; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Patients will also be given the opportunity to have serum samples stored for up to 10 years for future exploratory analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aspartylglucosaminuria (AGU) is a rare neurodegenerative lysosomal storage disease (LSD) characterized by developmental delay, psychomotor regression, worsening intellectual disability, gait disturbance and, ultimately, premature death, and has no available treatments.

The purpose of this study is to investigate the clinical characteristics and natural clinical progression of symptoms in individuals with AGU. This natural history study is important to better understand disease course to be able to determine clinically meaningful outcome measures for use in future clinical trials.

DETAILED DESCRIPTION:
Lysosomal storage disorders (LSDs) are a group of inherited metabolic diseases caused by a genetic mutation resulting in deficiency or absence of a critical enzyme, leading to the accumulation of toxic deposits in cells across multiple organ systems.

Aspartylglucosaminuria (AGU) is a rare, neurodegenerative, LSD, caused by a deficiency of the aspartylglucosaminidase (AGA) enzyme, which leads to toxic accumulation of aspartylglucosamine and subsequent cellular dysfunction. AGU has been most commonly reported in people of Finnish and Nordic descent, but is present across ethnicities and is typically misdiagnosed or undiagnosed.

Aspartylglucosaminuria (AGU) is characterized by developmental delay and intellectual disability that worsens with age. Early disease is characterized by increased frequency of bacterial ear infections, recurrent ear tube placement, intestinal dysfunction, disruptive sleep patterns, skeletal abnormalities, and gait disturbances, among others. Individuals progressively lose motor and cognitive skills, develop behavioral/emotional lability and their risk of seizures increases with age. People with AGU have a shortened life span.

No prospective natural history study for AGU has been reported. This study aims to prospectively investigate the natural history of AGU, and concurrently to identify potential outcome measures that could be used in future clinical trials. No investigational product will be provided in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of AGU based on clinical presentation and genetic testing (known or suspected pathogenic mutation in AGA gene).

Exclusion Criteria:

* Patients unable to travel to UT Southwestern Medical Center and Children's Health Dallas will not be enrolled in the prospective natural history study collecting standardized clinical data; however, with participant consent, medical records will be obtained, reviewed, and recorded in the natural history database over time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed genetic diagnosis of aspartylglucosaminuria.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Testing | 5 years
  Participants will undergo a standardized neuropsychological evaluation every 6-12 months, depending upon the assessments as follows:
  Global Cognitive: Leiter International Performance Scale, 3rd Ed, Reynolds Intellectual Assessment Scales, 2nd Ed, Mullen Scales of Early Learning
  Emotional: Aberrant Behavior Checklist, 2nd Ed, Behavior Assessment System for Children, 3rd Ed
  Behavioral functioning: Aberrant Behavior Checklist, 2nd Ed, Behavior Assessment System for Children, 3rd Ed
Ophthalmological Evaluation | 5 years
  Participants will undergo an ophthalmological assessment every 6 months to better characterize the involvement of the eye in AGU.
Visual Evoked Potential (VEP) | 5 years
  Participants will undergo a VEP test every 6 months to evaluate electrical signal transmission through the visual pathway from the retina to the visual cortex.
Brainstem Auditory Evoked Response (BAER) | 5 years
  Participants will undergo a BAER test every 6 months to evaluate electrical signal transmission from the 8th cranial nerve to the brainstem and the cortex in response to certain tones.
Magnetic Resonance Imaging (MRI)/Magnetic Resonance Spectroscopy (MRS) | 5 years
  An MRI scan of the brain will be performed annually to characterize the structural abnormalities associated with AGU. MRS will be performed on regions of interest in the brain.

SECONDARY OUTCOMES:
Adaptive functioning: Vineland Adaptive Behavior Scales, 3rd Ed | 5 years
  Participants will undergo a standardized neuropsychological evaluation every 6-12 months
Language: Expressive One-Word Picture Vocabulary Test, 4th Ed, Receptive One-Word Picture Vocabulary Test, 4th Ed, NEPSY, 2nd Ed | 5 years
  Participants will undergo a standardized neuropsychological evaluation every 6-12 months
Motor: NIH Toolbox Early Childhood Motor Battery or NIH Toolbox Motor Battery, 6 Minute Walk Test, Beery-Buktenica Development | 5 years
  Participants will undergo a standardized neuropsychological evaluation every 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elise Beausoleil, Study Director — Neurogene Inc.
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States